CLINICAL TRIAL: NCT03198793
Title: A Phase 2, Open-Label, Dose-Titrating Safety and Efficacy Study of QGC001 Administered Orally, Twice Daily, Over 8 Weeks in Hypertensive Overweight Subjects of Multiple Ethnic and Racial Groups in the United States
Brief Title: Novel Evaluation With QGC001 in Hypertensive Overweight Patients of Multiple Ethnic Origins
Acronym: NEW-HOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quantum Genomics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QGC001-2QG3
Record Dates: First submitted 2017-06-16; First posted 2017-06-26 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QGC001 (Experimental): Capsules of QGC001 250 mg
  Interventions: Drug: QGC001

INTERVENTIONS:
Drug: QGC001 — Twice daily (BID) administration of oral (PO) QGC001 (250 mg BID, 500 mg BID, and 500 mg BID + hydrochlorothiazide (HCTZ) 25 mg once daily [QD]) over 8 weeks.

SUMMARY:
Essential hypertension (HTN) is a disease that affects approximately 1 billion individuals worldwide. Despite the availability of effective and safe anti-hypertensive drugs, 65% of subjects diagnosed with HTN do not have their blood pressure (BP) controlled (<140/90 mmHg). The overall incidence of resistant HTN, (defined as requiring 3 or more anti-hypertensive drugs, including a diuretic, to control BP) is estimated to be 15% of the hypertensive population. Consequently, there is a pressing unmet medical need to develop new classes of anti-hypertensive drugs that act on alternative pathways and further control BP and the associated cardiovascular risks in subjects.

The prevalence of HTN in African Americans in the United States is among the highest in the world, and HTN is more common in African Americans than in Caucasians. One of the risk factors for HTN is sodium sensitivity. There is a higher association of HTN with sodium sensitivity in African American subjects and other racial/ethnic groups who are overweight/obese.

Effective agents to treat HTN in this high-risk population are clearly needed.

This study will be conducted in a hypertensive, overweight subject population of multiple ethnic origins in which QGC001 is likely, based on its mode of action, to demonstrate a significant anti-hypertensive effect.

DETAILED DESCRIPTION:
QGC001 is a prodrug of the specific and selective APA inhibitor, EC33, and is the prototype of a new class of centrally-acting anti-hypertensive agents called brain APA inhibitors. Inhibition of brain APA, which converts Ang II into Ang III, has emerged as a novel anti hypertensive treatment, as demonstrated in several experimental animal models. QGC001's anti-hypertensive effect is in part due to: 1) a decrease in arginine vasopressin release in the blood circulation, increasing diuresis, which reduces the size of body fluid compartment; and 2) a reduction in the sympathetic tone, leading to subsequent decreases in vascular resistances.

This study is an open-label, dose-titrating safety and efficacy study of QGC001 administered PO, BID, over 8 weeks in hypertensive overweight subjects of multiple ethnic and racial groups in the United States.

The primary objective of this study is to assess the effects of twice daily (BID) administration of oral (PO) QGC001 (250 mg BID, 500 mg BID, and 500 mg BID + hydrochlorothiazide (HCTZ) 25 mg once daily [QD]) on blood pressure (BP) over 8 weeks in hypertensive overweight/obese subjects of multiple races/ethnicities.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide signed written informed consent;
* Men and women greater than or equal to 18 years of age at Screening;
* Diagnosis of primary (essential) hypertension (HTN) for at least 3 months prior to Screening and have an office SBP:

  * Between 145 mmHg and 170 mmHg at Screening and are treatment-naïve; or
  * Between 130 mmHg and 150 mmHg at Screening and are treated with less than or equal to 2 anti hypertensive medications. Anti-hypertensive medications must be stable for greater than or equal to 8 weeks prior to Screening;
* SBP between 145 mmHg and 170 mmHg, inclusive, and DBP less than or equal to 105 mmHg at the Inclusion Visit after 2-week Run In Period;
* Body mass index between 25 kg/m2 and 45 kg/m2 with the ability to fit the ambulatory blood pressure monitoring (ABPM) cuff per the manufacturer;
* Subject must have a successful ABPM measurement prior to receiving the study drug.
* Women of childbearing potential and non-surgically sterile male subjects who are sexually active must agree to use an approved highly effective form of contraception from the time of informed consent until 30 days post-dose.
* Women of childbearing potential must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test result at the Inclusion Visit (Day 0).

Exclusion Criteria:

* Known or suspected secondary HTN (eg, renal artery stenosis, pheochromocytoma, Cushing's disease);
* Office SBP greater than or equal to 171 mmHg and/or office diastolic blood pressure (DBP) greater than or equal to 105 mmHg at the Inclusion Visit (Day 0) and confirmed by a second measurement (not on the same day), preferably within 1 day;
* Known hypertensive retinopathy (Keith-Wagener Grade 3 or Grade 4) and/or hypertensive encephalopathy;
* History of spontaneous or drug-induced angioedema;
* Clinically significant valvular heart disease or severe aortic stenosis;
* Subjects with symptomatic heart failure (New York Heart Association Class II to Class IV);
* History of acute coronary syndrome (non-ST elevation myocardial infarction, ST elevation myocardial infarction, and unstable angina pectoris), stroke, or transient ischemic attack within 6 months prior to Screening;
* Known history of malabsorption syndrome, or has undergone gastrointestinal surgery, including bariatric procedures, that induce chronic malabsorption, within 2 years of Screening;
* Treatment with anti-obesity drugs or procedures 3 months prior to Screening (ie, surgery, aggressive diet regimen, etc.), leading to unstable body weight;
* Female who is breast feeding, pregnant, or planning to become pregnant during the study period;
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years;
* Subject with an upper arm circumference that exceeds the upper circumference level (48.3 cm) of the cuff size of either the ABPM and/or office BP (OBP) measurement device used in the study;
* Night shift workers who routinely sleep during the daytime and/or whose work hours include midnight;
* Alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase >3 x upper limit of normal (ULN) or a total bilirubin greater than or equal to 2 x ULN (unless secondary to Gilbert's syndrome) at Screening or the Inclusion Visit (Day 0);
* Estimated glomerular filtration rate <45mL/min/1.73m2, as calculated using the Chronic Kidney Disease Epidemiology Collaboration formula at Screening or the Inclusion Visit (Day 0);
* History of any blood disorder, other than sickle cell trait, causing hemolysis or unstable red blood cells (eg, malaria, babesiosis, hemolytic anemia, thalassemia, sickle cell anemia);
* Subjects with type 1 diabetes mellitus;
* Subjects with type 2 diabetes mellitus who:

  * Are poorly controlled, defined as hemoglobin A1c >8% at Screening; or
  * Are taking short-acting insulin or sodium-glucose co transporter 2 inhibitors. Use of a stable dose (greater than or equal to 12 weeks prior to Screening) of medications listed in Appendix C is permitted;
* Routine or anticipated treatment with all systemic corticosteroids. Use of topical, inhaled, or nasal corticosteroids is permitted;
* Clinical evidence of thyroid disease, thyroid hormone therapy that is not stable greater than or equal to 4 weeks prior to Screening, or subjects with the following thyroid-stimulating hormone (TSH) levels at Screening:

  * For subjects on replacement therapy: TSH 0.75 to 1.5 x ULN; or
  * For subjects not on replacement therapy: TSH >1.5 x ULN;
* History of alcohol or drug abuse within the 3 months prior to Screening that would interfere with study participation or lead to decreased compliance to study procedures or study drug intake in the Investigator's opinion;
* Participation in another clinical study involving an investigational drug within 30 days prior to Screening, or plans to participate in another clinical study within 30 days of discontinuation of study drug;
* Any condition, in the opinion of the Investigator, that would interfere with study participation, may pose a risk to the subject, or would make study participation not in the best interest of the subject;
* Subjects with a life expectancy of less than 1 year per Investigator's discretion; or
* Any subject who, in the opinion of the Investigator, will not be able to follow the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Change in office systolic blood pressure from baseline to Week 8 (Day 56 Visit) | 8 weeks
  Office blood pressure will be taken at Day 0, Visit 3, Visit 4, Visit 4.1, and Visit 5 (Day 56).

SECONDARY OUTCOMES:
Change in office diastolic blood pressure from baseline to Week 8 (Day 56 Visit) | 8 weeks
  Office blood pressure will be taken at Day 0, Visit 3, Visit 4, Visit 4.1, and Visit 5 (Day 56).
Change in office systolic blood pressure and diastolic blood pressure from baseline to Week 4 (Day 28 Visit) | 4 weeks
  Office blood pressure will be taken at Day 0, Visit 3, Visit 4, Visit 4.1, and Visit 5 (Day 56).
Change in mean 24-hour ambulatory systolic blood pressure, diastolic blood pressure, and mean office blood pressure from baseline to Week 8 (Day 56 Visit) | 8 weeks
  Ambulatory blood pressure monitoring will be performed at Day 0 and Day 56.
Percentage of responders (defined as subjects with normalized office blood pressure, ie, less than or equal to 140-90 mmHg at Week 8 - Day 56 Visit) | 8 weeks
  Frequency and percentage of subjects who reach the level by the Week 8 (Day 56 Visit).
Predictive factors for responders at Week 8 (Day 56 Visit) | 8 weeks
  Identification of potential factors for responders, including baseline systolic blood pressure and diastolic blood pressure, gender, age, BMI, and others.

CONTACTS AND LOCATIONS:
Overall Officials: Keith C. Ferdinand, MD FACC, Study Chair — Tulane University SOM, New Orleans, LA 70112
Locations (1):
- Progressive Medical Research, Port Orange, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khosla J, Aronow WS, Frishman WH. Firibastat: An Oral First-in-Class Brain Aminopeptidase A Inhibitor for Systemic Hypertension. Cardiol Rev. 2022 Jan-Feb 01;30(1):50-55. doi: 10.1097/CRD.0000000000000360. PMID 33027067
- [Derived] Ferdinand KC, Harrison D, Johnson A. The NEW-HOPE study and emerging therapies for difficult-to-control and resistant hypertension. Prog Cardiovasc Dis. 2020 Jan-Feb;63(1):64-73. doi: 10.1016/j.pcad.2019.12.008. Epub 2020 Jan 8. PMID 31923435
- [Derived] Ferdinand KC, Balavoine F, Besse B, Black HR, Desbrandes S, Dittrich HC, Nesbitt SD. Efficacy and Safety of Firibastat, A First-in-Class Brain Aminopeptidase A Inhibitor, in Hypertensive Overweight Patients of Multiple Ethnic Origins. Circulation. 2019 Jul 9;140(2):138-146. doi: 10.1161/CIRCULATIONAHA.119.040070. Epub 2019 Apr 24. PMID 31014072